CLINICAL TRIAL: NCT05365230
Title: A Randomized Trial Evaluating Personalized vs Guideline-based Well Follow-up Strategies for Patients With Early-stage Breast Cancer (REaCT-Wellness)
Brief Title: A Randomized Trial Evaluating Personalized vs Guideline-based Well Follow-up Strategies for Patients With Early-stage Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REaCT-Wellness
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Well Follow-up; Follow-up Interval
MeSH Terms: conditions — Breast Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On-demand personalized follow-up care (Active Comparator): On-demand personalized follow-up care (on-demand access to a Wellness Beyond Cancer Program (WBCP) nurse and an annual follow-up by telephone with WBCP nurse following the patient's annual mammogram). Both groups of participants will have yearly mammograms (current standard of care) organized by their healthcare provider.
  Interventions: Other: On-demand personalized follow-up care
- Guideline-based follow-up care (Active Comparator): Guideline-based follow-up care (i.e. current standard of care). Both groups will have yearly mammograms (current standard of care) organized by their healthcare provider.
  Interventions: Other: Guideline-based follow-up care (standard of care)

INTERVENTIONS:
Other: On-demand personalized follow-up care — On-demand personalized follow-up care (on demand access to a WBCP nurse and an annual follow-up by telephone.
  Arms: On-demand personalized follow-up care
Other: Guideline-based follow-up care (standard of care) — Follow-up care based on current standard of care guidelines.
  Arms: Guideline-based follow-up care

SUMMARY:
After breast cancer patients complete the acute phase of their treatment (i.e. surgery, chemotherapy and/or radiation therapy), they are routinely followed in clinic every 3-6 months for several years. Multiple guideline recommendations exist with no consensus on the optimal follow-up schedule due to lack of randomized data to support any particular follow-up recommendation. Therefore the investigators propose a randomized trial evaluating personalized vs guideline-based well follow-up strategies for patients with early-stage breast cancer.

DETAILED DESCRIPTION:
After breast cancer patients complete the acute phase of their treatment (i.e. surgery, chemotherapy and/or radiation therapy), they are routinely followed in clinic every 3-6 months for several years. Multiple guideline recommendations exist with no consensus on the optimal follow-up schedule due to lack of randomized data to support any particular follow-up recommendation. The frequency of follow-up varies between and within different institutions. To date, no de-escalation strategy has appropriately evaluated patient reported outcomes such as quality of life or perception of care. There has been a growing body of evidence that de-intensification of follow-up is safe, effective and reduces costs for both patients and the health care system. Therefore the investigators propose a randomized trial evaluating personalized vs guideline-based well follow-up strategies for patients with early-stage breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Being referred to the Wellness Beyond Cancer Program (WBCP) for routine follow-up after completion of acute phase of treatment for invasive breast cancer

Exclusion Criteria:

* History of prior invasive breast cancer, recurrent brest cancer or metastatic breast cancer
* Currently receiving zoledronate, LHRH (Gonadotropin-releasing hormone) or abemaciclib

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Health-Related Quality of Life | 24 months after randomization
  Health-Related Quality of Life as determined by the Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire. The FACT-G is a 27-item questionnaire designed to measure four domains of Health related quality of life (HRQOL) in cancer patients: physical, social, emotional and functional well-being.

SECONDARY OUTCOMES:
Fear of recurrence | 24 months after randomization
  Fear of recurrence will be measured by the Functional Assessment of Cancer Therapy - Fear of Recurrence (FACT-FRQ) questionnaire. It consists of 3 questions suggested by David Cella at FACIT (Functional Assessment of Chronic Illness Therapy), that were adapted from Vickberg's Concerns about Recurrence (CARS) questionnaire.
Anxiety levels | 24 months after randomization
  Anxiety levels as determined by the Hospital Anxiety and Depression Scale (HADS) questionnaire. The HADS questionnaire measures anxiety and depression, which commonly coexist. It is comprised of seven questions for anxiety and seven questions for depression.
Treatment related toxicity concerns | 24 months after randomization
  Treatment related toxicity concerns as assessed using the Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) questionnaire. The FACT-ES questionnaire is a validated sub scale of the Functional Assessment of Chronic Illness Therapy (FACIT) measurement system. FACT-ES consists of 46 items on a 5 point Likert type scale ranging from 0 (not at all) to 4 (very much). It is designed to measure five domains of health: physical well-being, social/family well-being, emotional well-being, functional well being and endocrine symptom subscale.
Recurrence-free survival | 24 months after randomization
  Measured by the number of participants free of breast cancer recurrence after 24 months of follow-up.
Patient visits | 24 months after randomization
  Number of patient reported visits to different healthcare providers using a Patient Follow-up Questionnaire. The follow-up questionnaire consists of questions that assess the number of follow up visits a participant has had and also the type of healthcare provider the follow-up visits were with.
Cost-effectiveness | 24 months after randomization
  Incremental cost-effectiveness rations (cost per one quality-adjusted life year (QALY) gained.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Clemons, MD, Principal Investigator — The Ottawa Hospital Research Institute; John Hilton, MD, Principal Investigator — The Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Beltran-Bless AA, Alshamsan B, Alzahrani MJ, Hilton J, Baines KA, Samuel V, Pond GR, Vandermeer L, Clemons M, Larocque G. Regularly scheduled physical examinations and the detection of breast cancer recurrences. Breast. 2023 Jun;69:274-280. doi: 10.1016/j.breast.2023.03.004. Epub 2023 Mar 8. PMID 36922304
- [Background] Beltran-Bless AA, Larocque G, Brackstone M, Arnaout A, Caudrelier JM, Boone D, Fallah P, Ng T, Cross P, Alqahtani N, Hilton J, Vandermeer L, Pond G, Clemons M. The COVID-19 pandemic and its effects on follow-up of patients with early breast cancer: A patient survey. Breast Cancer Res Treat. 2024 Apr;204(3):531-538. doi: 10.1007/s10549-023-07232-3. Epub 2024 Jan 9. PMID 38194133
- [Background] Beltran-Bless AA, Larocque G, Arnaout A, Caudrelier JM, Hilton J, Alqahtani N, Vandermeer L, Pond G, Clemons M. Evolving strategies for the routine follow-up of patients with early breast cancer and the impact of COVID-19: a survey of healthcare providers. Support Care Cancer. 2025 Feb 27;33(3):232. doi: 10.1007/s00520-025-09205-2. PMID 40014172
- [Background] Beltran-Bless AA, Clemons M. How Frequently Should Patients with Breast Cancer Have Routine Follow-Up Visits? NEJM Evid. 2023 Aug;2(8):EVIDtt2300062. doi: 10.1056/EVIDtt2300062. Epub 2023 Jul 25. PMID 38320146
- [Background] Surujballi J, Shah H, Hutton B, Alzahrani M, Beltran-Bless AA, Shorr R, Larocque G, McGee S, Cole K, Ibrahim MFK, Fernandes R, Arnaout A, Stober C, Liu M, Sienkiewicz M, Saunders D, Vandermeer L, Clemons M. The COVID-19 pandemic: An opportunity to rethink and harmonise the frequency of follow-up visits for patients with early stage breast cancer. Cancer Treat Rev. 2021 Jun;97:102188. doi: 10.1016/j.ctrv.2021.102188. Epub 2021 Mar 23. PMID 33813329
- See also: The Rethinking Clinical Trials (REaCT) website — https://react.ohri.ca/